CLINICAL TRIAL: NCT03553966
Title: Impact of the Daily Use of Hydroxyapatite-toothpaste on the Occurrence of Enamel Caries in the Primary Dentition (ECIPDEN17)
Brief Title: Hydroxyapatite-toothpaste and Enamel Caries in the Primary Dentition
Acronym: ECIPDEN17
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Kurt Wolff GmbH & Co. KG (Industry)
Collaborators: Medical University of Bialystok (Other); Wuerzburg University Hospital (Other); Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Elzbieta Paszynska, DDS, PhD, Assoc. Prof.,, Dr. Kurt Wolff GmbH & Co. KG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dr. Kurt Wolff Group
Record Dates: First submitted 2018-04-23; First posted 2018-06-12 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Tooth Decay; Hydroxyapatite; Tooth Demineralization; Tooth Diseases
Keywords: Dental caries; Toothpaste; Fluoride; Hydroxyapatite
MeSH Terms: conditions — Dental Caries; Tooth Demineralization; Tooth Diseases

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, randomized, active-controlled parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tooth Brushing HAP+Restorative dentistry (Experimental): Arm Intervention: HA-Toothpaste Tooth Brushing HA Prophylactic cleaning of all teeth using a standardized electric tooth brush and a non-fluoridated toothpaste containing microcrystalline hydroxylapatite 3x daily over the duration of the study (336 days).
  Procedure: Tooth Brushing HA
  Interventions: Procedure: Prophylactic; Device: Restorative dentistry
- Tooth Brushing F+Restorative dentistry (Active Comparator): Cleaning teeth using a standardized electric tooth brush and a fluoridated tooth paste containing amino fluoride (500 ppm F-), (three times daily over the duration of the study (336 days).
  Intervention:
  Procedure: Tooth Brushing F 3x daily repeated cleaning of all teeth using a standardized electric tooth brush and a fluoridated toothpaste.
  Interventions: Procedure: Cleaning teeth; Device: Restorative dentistry

INTERVENTIONS:
Procedure: Prophylactic — Tooth Brushing HA 3x daily repeated cleaning of all teeth using a standardized electric tooth brush and a non-fluoridated tooth paste containing microcrystalline hydroxylapatite.
  Other Names: ECIPDEN17
  Arms: Tooth Brushing HAP+Restorative dentistry
Procedure: Cleaning teeth — Tooth Brushing F 3x daily repeated cleaning of all teeth using a standardized electric tooth brush and a fluoridated tooth paste.
  Other Names: ECIPDEN17
  Arms: Tooth Brushing F+Restorative dentistry
Device: Restorative dentistry — If in a subject a significant increase of carious lesions will be observed, her/his parents are informed about the necessity for further caries preventive measures (e.g. dietary changes, use of fluoride products, reduction of cariogenic microflora with chlorhexidine, xylitol chewing gum, etc.) and caries preventive treatment (removing caries and placing a restoration) by the study centers is offered.

SUMMARY:
This multicenter, non-inferiority trial randomized, double-blind, active controlled parallel group study evaluates the hypothesis that the home regular use of a toothpaste containing microcrystalline hydroxylapatite (HAP) (test toothpaste) provides a caries preventive effect in caries-active children with primary dentition age 3-6 which is comparable to the caries preventive effect provided by the regular use of a fluoridated tooth paste (F) (control toothpaste) over observation periods of max. 336 days. Caries development will be assessed according to the clinical criteria of the International Caries Detection and Assessment System (ICDAS).

Condition or disease:

Intervention Procedure: Tooth Brushing HAP or Procedure: Tooth Brushing F

DETAILED DESCRIPTION:
According to the criteria of evidence based medicine the use of fluoridated tooth paste (as well as fluoridated mouth rinses) with the exception of dietary control, are the only proven measures for the prevention of dental caries. Regular tooth brushing with a fluoridated toothpaste represents the golden standard of oral care also in the primary dentition established by numerous clinical studies.

Fluorides are widely used for caries prevention. However, particularly in children and adolescents the dosage of fluorides in oral care products must be carefully monitored, as chronic overdosing of fluoride may negatively interfere with the mineralization of dentin and enamel (fluorosis). Therefore the acceptable concentration of fluorides in oral care products is limited and regulated by the European Regulation (EC) No. 12223/2009 on cosmetic products:

REGULATION (EC) No 1223/2009 OF THE EUROPEAN PARLIAMENT AND OF THE COUNCIL of 30 November 2009 on cosmetic products "For any toothpaste containing 0.1 to 0.15% fluoride unless it is already labelled as contra-indicated for children (e.g. 'for adult use only') the following labelling is obligatory: 'Children of 6 years and younger: Use a pea sized amount for supervised brushing to minimize swallowing. In case of intake of fluoride from other sources consult a dentist or doctor'" Toothpastes suitable for children up to six years may only contain 500 ppm due to the risk of increased fluoride uptake by swallowing the toothpaste. However, such reduced fluoride contents may also reduce the caries prophylactic efficacy of the toothpaste particularly in highly caries-active individuals (Walsh et al. 2010). Therefore, especially for children there is a need for efficacious alternative (non-toxic) caries-preventing agents.

Target Question:

Does the regular use of a fluoride-free, microcrystalline hydroxyapatite (HAP) - containing test toothpaste have a non-inferior impact on the incidence of enamel caries in the primary dentition compared to the regular use of a fluoridated control toothpaste with proven caries preventive efficacy? The aim of this clinical trial is to assess in cohorts of caries-active children with primary teeth whether daily tooth brushing at home over observation periods of max. 336 days with a hydroxyapatite-containing toothpaste (test toothpaste) provides a protection from enamel caries development which is not inferior to the protection when brushing with a fluoridated toothpaste (control toothpaste).

Material and Methods Subjects

Study subjects will be recruited from a target population of caries-active children with primary teeth aged ≥ 3 to 6 years. The target population we be stratified according to the number of filled molars:

There will be 2 strata:

Stratum A: Children with high risk of caries development. Either 1-2 filled molars or 1-2 molars with at least ICDAS 4, which will be dentally treated. Thus, 6-7 enamel surfaces can be assessed.

Stratum B: Children with very high risk of caries development. Either 3-4 filled molars or 3-4 molars with at least ICDAS 4, which will be dentally treated. Thus, 4-5 enamel surfaces can be assessed.

Number of test centers and subjects The trial will be performed at three test centers (Poznan, Bialystok, Regensburg) Total number of subjects to be enrolled: n=200

Methods Test intervention: Oral hygiene instruction and regular domestic application of the test toothpaste (3x daily over a period of 336 days); also during weekends and holidays Reference (control) intervention: Oral hygiene instruction and regular domestic application of the fluoridated (reference) toothpaste (3x daily over a period of 336 days); also during weekends and holidays (The reference intervention corresponds to the established scientific standard for the prevention of enamel caries in primary teeth).

The following parameters will be evaluated each three months:

* caries development will be assessed according to the clinical criteria of the International Caries Detection and Assessment System (ICDAS), (Ismail et al 2007).
* changes in the coverage of the assessed primary molars with bacterial plaque according to the criteria of the Plaque Control Record.
* changes in the status of gingival health in the gingiva of the assessed primary molars according to the criteria of the Modified Gingival Index.

ELIGIBILITY:
Inclusion Criteria:

* age 3-6 years
* complete set of fully erupted primary molars (teeth 55, 54, 64, 65, 75, 74, 84, 85)
* presence of a caries restoration (filling) on a minimum of 1 primary molar
* minimum of 4 primary molars without a restoration or fissure sealing

Exclusion Criteria:

* untreated caries lesions of ICDAS code 3-6
* known hypersensitivity to one of the ingredients of the toothpastes to be tested
* systemic disorders interfering with salivary function or flow
* regular medication intake interfering with salivary function or flow
* need for antibiotic prophylaxis during dental treatments
* participation in any other clinical study within the past 3 months or ongoing
* lack of intellectual or physical ability to conduct the study properly
* any other reason that, in the opinion of the investigator, disqualifies the subject from participating in the study

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of study subjects experiencing new enamel caries lesions (≥ ICDAS code 1) | 336 days
  Percentage of study subjects experiencing the new development of at least one enamel caries lesions ≥ ICDAS code 1 or the progression of an existing enamel caries lesion by at least one ICDAS code on any of the evaluated primary molars during the observation period of 336 days.
  Reference: ICDAS II code (International Caries Detection and Assessment System; ICDAS); Ismail et al. 2007.

SECONDARY OUTCOMES:
Gingival Inflammation using the Gingival Index | 336 days
  Changes in the status of gingival health in the gingiva of the assessed primary molars according to the criteria of the Modified Gingival Index..
Plaque Coverage using the Plaque Control Record | 336 days
  Changes in the coverage of the assessed primary molars with bacterial plaque according to the criteria of the Plaque Control Record.
Percentage of study subjects experiencing new enamel caries lesions (≥ ICDAS code 2) | 336 day
  Percentage of study subjects experiencing the new development of at least one enamel caries lesions ≥ ICDAS code 2 during the observation period (336 days).

CONTACTS AND LOCATIONS:
Overall Officials: Elzbieta Paszynska, Assoc. Prof., Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Department of Integrated Dentistry, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No
we do not plan any individual participant data available data to other researchers

REFERENCES:
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012 Dec 26;308(24):2594-604. doi: 10.1001/jama.2012.87802. PMID 23268518
- [Background] Walsh T, Worthington HV, Glenny AM, Appelbe P, Marinho VC, Shi X. Fluoride toothpastes of different concentrations for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD007868. doi: 10.1002/14651858.CD007868.pub2. PMID 20091655
- [Background] REGULATION (EC) No 1223/2009 OF THE EUROPEAN PARLIAMENT AND OF THE COUNCIL of 30 November 2009 on cosmetic products. (2009).
- [Background] Kensche A, Holder C, Basche S, Tahan N, Hannig C, Hannig M. Efficacy of a mouthrinse based on hydroxyapatite to reduce initial bacterial colonisation in situ. Arch Oral Biol. 2017 Aug;80:18-26. doi: 10.1016/j.archoralbio.2017.03.013. Epub 2017 Mar 23. PMID 28364672
- [Result] Hiller KA, Buchalla W, Grillmeier I, Neubauer C, Schmalz G. In vitro effects of hydroxyapatite containing toothpastes on dentin permeability after multiple applications and ageing. Sci Rep. 2018 Mar 20;8(1):4888. doi: 10.1038/s41598-018-22764-1. PMID 29559639
- [Result] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Result] Luz PB, Stringhini CH, Otto BR, Port AL, Zaleski V, Oliveira RS, Pereira JT, Lussi A, Rodrigues JA. Performance of undergraduate dental students on ICDAS clinical caries detection after different learning strategies. Eur J Dent Educ. 2015 Nov;19(4):235-41. doi: 10.1111/eje.12131. Epub 2014 Dec 12. PMID 25495379
- [Result] Loe H. Mechanical and chemical control of dental plaque. J Clin Periodontol. 1979 Dec;6(7):32-6. doi: 10.1111/j.1600-051x.1979.tb02116.x. No abstract available. PMID 295293
- [Result] Milsom KM, Blinkhorn AS, Tickle M. The incidence of dental caries in the primary molar teeth of young children receiving National Health Service funded dental care in practices in the North West of England. Br Dent J. 2008 Oct 11;205(7):E14; discussion 384-5. doi: 10.1038/sj.bdj.2008.582. PMID 18849940
- [Result] World Medical Association: Declaration of Helsinki. Recommendations guiding medical physi-cians in biomedical research involving human subjects, 59th WMA General Assembly, Seoul, October, 2008
- [Result] International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) adopts Consolidated Guideline on Good Clinical Practice in the Conduct of Clinical Trials on Medicinal Products for Human Use. Int Dig Health Legis. 1997;48(2):231-4. No abstract available. PMID 11656783
- [Result] Harks I, Jockel-Schneider Y, Schlagenhauf U, May TW, Gravemeier M, Prior K, Petersilka G, Ehmke B. Impact of the Daily Use of a Microcrystal Hydroxyapatite Dentifrice on De Novo Plaque Formation and Clinical/Microbiological Parameters of Periodontal Health. A Randomized Trial. PLoS One. 2016 Jul 28;11(7):e0160142. doi: 10.1371/journal.pone.0160142. eCollection 2016. PMID 27467683
- [Result] Lelli M, Putignano A, Marchetti M, Foltran I, Mangani F, Procaccini M, Roveri N, Orsini G. Remineralization and repair of enamel surface by biomimetic Zn-carbonate hydroxyapatite containing toothpaste: a comparative in vivo study. Front Physiol. 2014 Sep 5;5:333. doi: 10.3389/fphys.2014.00333. eCollection 2014. PMID 25249980
- [Derived] Paszynska E, Pawinska M, Gawriolek M, Kaminska I, Otulakowska-Skrzynska J, Marczuk-Kolada G, Rzatowski S, Sokolowska K, Olszewska A, Schlagenhauf U, May TW, Amaechi BT, Luczaj-Cepowicz E. Impact of a toothpaste with microcrystalline hydroxyapatite on the occurrence of early childhood caries: a 1-year randomized clinical trial. Sci Rep. 2021 Jan 29;11(1):2650. doi: 10.1038/s41598-021-81112-y. PMID 33514787